CLINICAL TRIAL: NCT03752957
Title: Wide-Awake Local Anesthesia No Tourniquet Versus. Local/General Anesthesia for Flexor Tendon Repair
Brief Title: Wide-Awake Local Anesthesia For Flexor Tendon Repair
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Slah Eldin Koriem, Assistant Lecturer, Assiut University
Other Study IDs: WideAwake Flexor Tendon Repair
Record Dates: First submitted 2018-11-05; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Flexor Tendon Injury
Keywords: Wide-Awake Local Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary repair for flexor tendon lacerations remain the standard of care. However, despite recent advances in knowledge of tendon healing, suture material, and post-operative protocols, outcomes have been reported as fair or poor in 7-20% of patients. Complications encountered include adhesion formation, development of joint contractures, tendon rupture, triggering, bow stringing and quadriplegia. Tendon surgery is unique because it should ensure tendon gliding after surgery Tendon surgery now can be performed under local anesthesia without tourniquet, by injecting epinephrine mixed with lidocaine, to achieve vasoconstriction in the area of surgery. This method allows the tendon to move actively during surgery to test tendon function intraoperatively and to ensure the tendon is properly repaired before leaving the operating table.

Wide awake hand surgery is well described by its other name, WALANT which stands for wide awake local anaesthesia no tourniquet. The only two medications most patients are given for wide awake hand surgery are Lidocaine for anaesthesia and epinephrine for haemostasis. In the period before 1950, the belief developed among surgeons that epinephrine causes finger necrosis .The source of the epinephrine myth stemmed from the use of procaine (Novocaine). It was the only safely injectable local anaesthetic until the introduction of Lidocaine in 1948. More fingers died from procaine injection alone than from procaine plus epinephrine injection .no lost finger no case require phentolamine in many studies.

DETAILED DESCRIPTION:
Primary repair for flexor tendon lacerations remain the standard of care. However, despite recent advances in knowledge of tendon healing, suture material, and post-operative protocols, outcomes have been reported as fair or poor in 7-20% of patients. Complications encountered include adhesion formation, development of joint contractures, tendon rupture, triggering, bowstringing and quadrigia. Tendon surgery is unique because it should ensure tendon gliding after surgery It has been a standard practice to obtain local or general anesthesia and apply a tourniquet to perform tendon surgery. However, this practice has been changed in recent years...

Tendon surgery now can be performed under local anesthesia without tourniquet, by injecting epinephrine mixed with lidocaine, to achieve vasoconstriction in the area of surgery. This method allows the tendon to move actively during surgery to test tendon function intraoperatively and to ensure the tendon is properly repaired before leaving the operating table.

The surgeon can inspect for bunching, gapping, and triggering of the repair site in an active fashion. Thus, an opportunity is available to revise the repair, trim or add extra sutures, revise pulley reconstruction, or de-bulk tendons before wound closure Wide awake hand surgery is well described by its other name, WALANT which stands for wide awake local anaesthesia no tourniquet. The only two medications most patients are given for wide awake hand surgery are Lidocaine for anaesthesia and epinephrine for haemostasis. In the period before 1950, the belief developed among surgeons that epinephrine causes finger necrosis .The source of the epinephrine myth stemmed from the use of procaine (Novocaine).8 It was the only safely injectable local anaesthetic until the introduction of Lidocaine in 1948. More fingers died from procaine injection alone than from procaine plus epinephrine injection .no lost finger no case require phentolamine in many studies.The "smoking gun" paper that established that procaine was the actual cause of finger deaths published in the Journal of the American Medical Association that found batches of procaine with a pH of 1 destined for injection into humans.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 acute single or multiple digit complete flexor tendon lacerations in zones I or II

Exclusion Criteria:

* gross wound contamination
* segmental tendon loss
* associated finger fractures
* complex or multisystem injuries
* complex or multisystem injuries
* mangled hand injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Assiut University Hospital , microsurgery unit
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
post operative complication rate | average 2 months
  Infection requiring antibiotics, tendon rupture, stiffness or contracture requiring tenolysis

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abdula ELgamal, Study Chair — Assiut University; Amr Elsaid Ali, Study Chair — Assiut University; Mohamed Mostafa Kotb, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No